CLINICAL TRIAL: NCT04063566
Title: ReIMAGINE Prostate Cancer Screening - Inviting Men for Prostate Cancer Screening Using MRI
Brief Title: ReIMAGINE Prostate Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Medical Research Council (Other Government); Cancer Research UK (Other); Imperial College London (Other); King's College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 123874
Record Dates: First submitted 2019-08-15; First posted 2019-08-21 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Prostate Cancer Screening; Prostate Cancer
Keywords: Prostate Cancer; MRI; PSA
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Spectroscopy; Prostate-Specific Antigen

STUDY DESIGN:
Intervention Model Description: Single site screening study to assess the feasibility of MRI as a screening tool for prostate care and determine the prevalence of MRI defined suspicious lesions and cancer in men across a spectrum of PSA results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Total cohort (Other): The study will consist of one group, one arm, all receiving the same screening procedures.
  Interventions: Procedure: Magnetic Resonance Imaging (MRI); Procedure: Prostate-specific antigen (PSA) test

INTERVENTIONS:
Procedure: Magnetic Resonance Imaging (MRI) — Prostate cancer screening MRI
Procedure: Prostate-specific antigen (PSA) test — Blood test for PSA levels

SUMMARY:
Single site study to assess the feasibility of prostate cancer screening using an invitation for a prostate MRI scan via GP practices. This feasibility study will assess the acceptability of an MRI as a prostate cancer screening assessment and assess the prevalence of MRI defined suspicious lesions and cancer in men across a spectrum of PSA results.

DETAILED DESCRIPTION:
ReIMAGINE Prostate cancer screening is a single site screening study to assess the feasibility of MRI as a screening tool for prostate care and determine the prevalence of MRI defined suspicious lesions and cancer in men across a spectrum of PSA results.

Men with no previous prostate cancer diagnosis, but deemed suitable based on age will be identified through general practitioner (GP) practices who will act as participant identification centres (PIC's). Potential participants will be identified through screening of existing patient databases at multiple London GP surgeries participating in the study, and randomly selected for invitation. The ReIMAGINE study team will link with London cancer networks and Noclor research support (https://www.noclor.nhs.uk/) who will make first contact with potentially eligible men.

A personalised invitation letter from each man's own GP will be sent to him. Invitation letters will be sent in batches so to limit the time between the invitation and their study visit. Batched invitations will be prepared using an iterative process so to allow the study team to assess uptake rates and limit the gap between invitation and study visits.

Invitation letters will include contact details for the ReIMAGINE study team who will coordinate bookings for research visits for all responders.

All consented men will have a blood test for PSA and a screening MRI scan. This will take a maximum of 20 minutes, and will include T2, diffusion and research specific sequences.

Two radiologists will report the MRI blinded to the PSA result, with a third reviewer when there is disagreement between reporters. Men in whom a suspicious lesion is seen (MRI screen positive) or who have a suspicious PSA density (>0.12ng/ml) will be recommended to have an National Health Service (NHS) referral for suspected prostate cancer as per National Institute for Health and Care Excellence (NICE) guidelines.

Screen negative men will at this point exit the study. Screen positive men will be followed up to gather data from any investigations (mpMRI +/- prostate biopsy) that may occur as a result of the NHS referral. No formal visits will be required to collect this data. Participant consent will be sought to approach GP or other secondary care centre.

ELIGIBILITY:
Inclusion Criteria:

1. Men aged 50-75
2. No prior prostate cancer diagnosis / treatment
3. Willing and able to provide written informed consent.

Exclusion Criteria:

1. Contraindication for MRI scanning (as assessed by the MRI safety questionnaire of the PET/MRI department) which includes but is not limited to: Intracranial aneurysm clips or other metallic objects; Intra-orbital metal fragments that have not been removed; Pacemakers or other implanted cardiac rhythm management devices and non-MRI compatible heart valves; Inner ear implants; and History of claustrophobia
2. Men who require assisted living e.g. care home living
3. Dementia or other neurological condition meaning participant lacks the capacity to consent.

Ages: 50 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 309 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
The acceptance rate of an invitation for a screening prostate MRI in men who have not had a prostate cancer diagnosis | 3 years
  Proportion of men who accept the invitation for prostate screening
The prevalence of MRI defined suspicious lesions in men accepting a screening invitation | 3 years
  The prevalence of MRI defined suspicious lesions in men accepting a screening invitation
Presence of cancer in men who have biopsy as a result of their MRI findings | 3 years
  The prevalence of men being diagnosed with prostate cancer who have biopsy as a result of their MRI findings

SECONDARY OUTCOMES:
The proportion of men ineligible due to prior prostate cancer diagnosis | 3 years
  The proportion of men ineligible due to prior prostate cancer diagnosis
The proportion of men who screen negative on MRI | 3 years
  The proportion of men who screen negative on MRI
The proportion of men who screen negative on PSA density | 3 years
  The proportion of men who screen negative on PSA density
The proportion of men who screen positive on MRI alone | 3 years
  The proportion of men who screen positive on MRI alone
The proportion of men who screen positive on PSA density alone | 3 years
  The proportion of men who screen positive on PSA density alone

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Moore, FRCS, Principal Investigator — univeristy college london
Locations (1):
- University College London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moore CM, Frangou E, McCartan N, Santaolalla A, Kopcke D, Brembilla G, Hadley J, Giganti F, Marsden T, Van Hemelrijck M, Gong F, Freeman A, Haider A, Tuck S, Pashayan N, Callender T, Green S, Brown LC, Punwani S, Emberton M. Prevalence of MRI lesions in men responding to a GP-led invitation for a prostate health check: a prospective cohort study. BMJ Oncol. 2023 Aug 21;2(1):e000057. doi: 10.1136/bmjonc-2023-000057. eCollection 2023. PMID 39886504
- [Derived] Marsden T, Lomas DJ, McCartan N, Hadley J, Tuck S, Brown L, Haire A, Moss CL, Green S, Van Hemelrijck M, Coolen T, Santaolalla A, Isaac E, Brembilla G, Kopcke D, Giganti F, Sidhu H, Punwani S, Emberton M, Moore CM; ReIMAGINE Study Group. ReIMAGINE Prostate Cancer Screening Study: protocol for a single-centre feasibility study inviting men for prostate cancer screening using MRI. BMJ Open. 2021 Sep 30;11(9):e048144. doi: 10.1136/bmjopen-2020-048144. PMID 34593491
- [Derived] Wurnschimmel C, Kachanov M, Wenzel M, Mandel P, Karakiewicz PI, Maurer T, Steuber T, Tilki D, Graefen M, Budaus L. Twenty-year trends in prostate cancer stage and grade migration in a large contemporary german radical prostatectomy cohort. Prostate. 2021 Sep;81(12):849-856. doi: 10.1002/pros.24181. Epub 2021 Jun 10. PMID 34110033
- [Derived] Marsden T, McCartan N, Hadley J, Tuck S, Brown L, Haire AJ, Moss CL, Green S, Van Hemelrijck M, Coolen T, Santaolalla A, Isaac E, Brembilla G, Kopcke D, Giganti F, Sidhu H, Punwani S, Emberton M, Moore CM; ReIMAGINE Study Group. Update from the ReIMAGINE Prostate Cancer Screening Study NCT04063566: Inviting Men for Prostate Cancer Screening Using Magnetic Resonance Imaging. Eur Urol Focus. 2021 May;7(3):503-505. doi: 10.1016/j.euf.2021.03.027. Epub 2021 Apr 23. PMID 33896710